CLINICAL TRIAL: NCT02649296
Title: Effect of Skanlab Regarding Knee Arthrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo Metropolitan University (Other)
Responsible Party: Principal Investigator, Hilde Sylliaas, Ass Prof, Oslo Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: Skanlab
Record Dates: First submitted 2015-10-29; First posted 2016-01-07 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Arthrosis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment with Skanlab Bodywave (Other): Treatment with Skanlab Bodywave twice a week for four weeks at the affected knee.
  Interventions: Other: Skanlab bodywave
- No treatment (No Intervention): Treatment with Skanlab Bodywave without function twice a week for four weeks.

INTERVENTIONS:
Other: Skanlab bodywave — The intervention will be done twice a week
  Arms: Treatment with Skanlab Bodywave

SUMMARY:
The purpose is to find out the effect of Skanlab at knee arthrosis.

DETAILED DESCRIPTION:
The patients diagnosed with knee arthrosis will be treated With Skanlab twice a week for four weeks.

ELIGIBILITY:
Inclusion Criteria:

* knee arthrosis in one or both legs

Exclusion Criteria:

* Pacemaker
* infusion pump
* cancer
* diabetes
* pregnancy
* blood clots
* bacteriological inflammation
* reduced sensitivity in the treatment area.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-01 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) | 15 months
  changes in pain

CONTACTS AND LOCATIONS:
Overall Officials: Trine Haugen, Prof, Study Director — Oslo and Akershus university college of applied science
Locations (1):
- Oslo and Akershus University college of applied science, Oslo, Norway, Norway